CLINICAL TRIAL: NCT00004486
Title: Randomized Study of Fluoxetine in Children and Adolescents With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 199/14266; MTS-FDR001520; MTS-GCO-96-713
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-12

CONDITIONS: Autism
Keywords: autism; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Autistic Disorder; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Fluoxetine

INTERVENTIONS:
Drug: fluoxetine

SUMMARY:
OBJECTIVES: I. Evaluate the efficacy of fluoxetine on social and language deficits, global severity and compulsive dimensions of children and adolescents with autism.

II. Assess the effectiveness of this treatment regimen on neurocognitive deficits in this patient population.

III. Compare the baseline compulsive severity and treatment outcome in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, crossover study. All patients receive oral placebo daily during week 0.

Patients are randomized to receive either oral fluoxetine or oral placebo daily on weeks 1-8. Patients then crossover to receive treatment on the other arm during weeks 12-20.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Meets diagnostic criteria for autism

--Prior/Concurrent Therapy--

Other:

* At least 3 months since prior electroconvulsive therapy
* At least 1 month since prior investigational drugs or treatment with any drug known to cause major organ toxicity
* At least 2 weeks since prior monoamine oxidase inhibitors
* At least 6 weeks since prior long acting phenothiazines
* At least 1 week since prior other psychotropic drugs
* No prior fluoxetine of 20 mg/day for 6 weeks
* At least 6 weeks since prior fluoxetine
* No concurrent use of terfenadine (Seldane) or astemizole (Hismanal)
* No concurrent electroconvulsive therapy or other psychotropic drugs (unless otherwise permitted)
* Prior participation in another serotonin reuptake inhibitor trial allowed

--Patient Characteristics--

Hematopoietic: No significant hematopoietic disease

Hepatic: No prior or concurrent liver disease

Renal: No prior or concurrent kidney disease

Cardiovascular:

* No significant cardiovascular disease
* No abnormal EKG

Neurological:

* No prior seizure disorder or high risk development of seizures
* No prior cerebrovascular disease
* No prior brain trauma

Other:

* Not pregnant or nursing
* Negative pregnancy test
* No unstable major medical illness or systemic disease
* No moderate or severe mental retardation and motor deficits (IQ less than 50)
* No family history of bipolar disorder
* No prior or concurrent other mental disorders (e.g., schizophrenia, schizoaffective, organic, or bipolar disorders)
* No significant autoaggressive behavior or serious suicidal risk
* No prior or concurrent gastrointestinal conditions
* No unstable endocrine disease (e.g., hypo or hyperthyroidism)
* No prior or concurrent malignancy
* Must be able to tolerate tapering of psychoactive medication
* No history of hypersensitivity or severe side effects to fluoxetine or other serotonin reuptake inhibitors
* No history of severe personality disorder or noncompliance

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45
Dates: Start 1998-09; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - New York University Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York

REFERENCES:
- [Result] Hollander E, Phillips A, Chaplin W, Zagursky K, Novotny S, Wasserman S, Iyengar R. A placebo controlled crossover trial of liquid fluoxetine on repetitive behaviors in childhood and adolescent autism. Neuropsychopharmacology. 2005 Mar;30(3):582-9. doi: 10.1038/sj.npp.1300627. PMID 15602505
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711